CLINICAL TRIAL: NCT02339402
Title: NON-INVASIVE PRENATAL TESTING (NIPT) OF FETAL SINGLE-GENE DISORDERS IN MATERNAL BLOOD
Brief Title: Non Invasive Prenatal Testing (NIPT) of Single-gene Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL48304/METC azM/UM 14-02-012
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Hereditary Disease
Keywords: Cystic fibrosis, Myotonic dystrophy, Noonan, Huntingtons
MeSH Terms: conditions — Genetic Diseases, Inborn; Cystic Fibrosis; Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Foetal DNA is isolated from the blood of pregnant women and their partners
Oversight: Data Monitoring Committee: No

SUMMARY:
Developing a new non-invasive prenatal test for single gene disorders from cell free fetal DNA, retrieved from the mothers blood.

DETAILED DESCRIPTION:
Rationale: Conventional prenatal diagnosis (PND) for single-gene disorders requires invasive procedures, either chorionic villus sampling between 11 and 14 weeks gestation or amniocentesis after 15 weeks. Although these approaches to obtain foetal DNA currently provide the golden standard for PND, the invasive procedures carry a risk of miscarriage of 0.5-1%. A reliable non-invasive alternative has long been sought. Circulating cell-free foetal (cff) nucleic acids (DNA and RNA), which are present in maternal blood during pregnancy, can be used for non-invasive prenatal testing (NIPT). NIPT for some chromosomal anomalies (trisomy 21, 13, 18) is now validated. NIPT for other chromosomal anomalies is still under development. NIPT of single-gene disorders is technically very challenging, due to the predominance of maternal DNA sequences, Some small studies have shown that a very limited number of monogenic genetic disorders can currently be diagnosed in maternal blood. In general de novo mutations in the foetus and paternally transmitted disorders are less difficult to diagnose than maternally transmitted disorders.

In this study, the investigators aim to develop non-invasive targeted molecular analysis using cell free fetal (cff) DNA and cff RNA for single-gene disorders, in pregnant women referred to the departments of Clinical Genetics of Maastricht University Medical Centre (MUMC+) and Radboud University Medical Centre (RUMC) for conventional PND. The investigators will contribute to literature by confirming earlier published results, and by adding other single-gene disorders or mutations to the list of disorders for which the possibility of the use of cff DNA will be examined.

Objective: Developing targeted non-invasive prenatal analysis for single-gene disorders using cff DNA and RNA in maternal plasma.

Study design: This study is a proof of concept study in which we aim to demonstrate that molecular analysis can indicate the presence or absence of (a) mutant allele(s) in maternal plasma.

Study population: Pregnant women (≥18y) referred to the Department of Clinical Genetics of MUMC+ or RadboudUMC for conventional PND, for one of the following reasons:

* The fetus is at high risk of having inherited a dominant or recessive disorder of his/her affected parent(s).
* The fetus at risk of having a de novo disorder on the basis of ultrasonography findings.

Main study endpoints: Does targeted molecular analysis of cff DNA and RNA indicate

1. the presence or absence of (a) mutant allele(s) in maternal plasma
2. the presence of a sufficient concentration of foetal nucleic acids in the maternal plasma to reliably diagnose the monogenic disorder Nature and extent of the burden and risks associated with participation and benefit: minimal burden: one moment of blood sampling for the pregnant woman and her partner. In most cases the blood sampling will be combined with regular blood sampling. Benefit: no benefit for this pregnancy as in the study phase the result of the invasive prenatal test is leading.

ELIGIBILITY:
Inclusion Criteria:

* the pregnant woman is scheduled for or has recently undergone invasive prenatal testing (regular care) because of one of the following reasons:

  * the fetus is at high risk of a having inherited a single-gene disorder from his/her affected parent(s).
  * the fetus is at risk of having a de dominant novo disorder on the basis of ultrasonography findings.
* the pregnant woman is 18 years or older
* the pregnant woman has sufficient understanding of Dutch language and is able to give informed consent

Exclusion Criteria:

* if in the opinion of the treating physician psychological distress is so severe that asking for participation is not safe
* the pregnant woman is treated for a malignancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women and their partner (≥18y) that undergo an invasive procedure for prenatal genetic diagnosis in the MUMC+ of RUMC for one of the following indications:
  * fetus at high risk of having inherited a dominant or recessive disorder of his/her affected parent(s) or
  * fetus at risk of having a de novo disorder on the basis of ultrasonography findings.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Development of a targeted molecular test (mostly standard PCR or real-time PCR) for non-invasive prenatal testing of single-gene disorders. | 2014-2016
  Main aims are to
  1. demonstrate the presence or absence of (a) mutant allele(s) in maternal plasma
  2. examine if there is a sufficient concentration of fetal nucleic acids in the maternal plasma to reliably diagnose the monogenic disorder

CONTACTS AND LOCATIONS:
Overall Officials: Christine de Die, MD PhD, Principal Investigator — Maastricht UMC
Locations (2):
- Netherlands (2):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastricht UMC, Maastricht